CLINICAL TRIAL: NCT03747991
Title: Effect of Histamine-2 Receptor Antagonists on the Microbiome of Full Term Infants
Brief Title: How Reflux Medications Affect the Microbiome of Infants
Status: Completed | Type: Observational
Sponsor: Nemours Children's Clinic (Other)
Responsible Party: Principal Investigator, Matthew Di Guglielmo, Chief, Division of General Academic Pediatrics, Nemours Children's Clinic
Other Study IDs: 1231469
Record Dates: First submitted 2018-11-16; First posted 2018-11-20 (Actual); Last update posted 2024-06-12 (Actual); Status verified 2024-06

CONDITIONS: GERD; Dysbiosis
Keywords: Infant GERD; H2RA medication
MeSH Terms: conditions — Gastroesophageal Reflux; Dysbiosis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Control Infants: Infants ages 2 months to 12 months who are not on H2RA medication.
- Treated Infants: Infants ages 2 months to 12 months who are taking H2RA medication.

SUMMARY:
The changes in the organisms making up the gut microbiota in infants who are taking anti-acid reflux medications (histamine 2 receptor antagonists) as compared to infants who are not taking these medications is not well-studied or understood. Whether these medications change the gut microbiota and microbiome, and what that change may imply for children on these medications, is the focus of this study.

DETAILED DESCRIPTION:
Gut microbiota dysbiosis is associated with diseases ranging from localized gastrointestinal disorders to neurologic, respiratory, metabolic, hepatic, and cardiovascular illnesses. The microbial colonization of the infant gut is known to play a key role in immunologic and metabolic pathways impacting on human health. Disruptions during the complex process of microbial colonization have been shown to increase disease susceptibility during life. A variety of factors are known to influence the gut microbiota, including mode of delivery of neonate, host genetic factors, hose immune response, diet, xenobiotics and other drugs, infections, and environmental microbial exposures.

The diagnosis of gastroesophageal reflux disease in the infant population has increased during the past two decades. Acid suppression medications are used commonly in infants for gastroesophageal reflux disease and other acid-related conditions despite little evidence of their efficacy. Multiple studies have shown adverse effects in pediatric patients using either proton pump inhibitors or H2 receptor antagonists, the two classes of acid suppression medications that are most frequently used in children. Some of these adverse effects may result from alterations in the microbiome caused by these medications. Prior studies have demonstrated significant changes in microbial composition of both gastric and intestinal microbiota with proton pump inhibitor use (5), but to the investigators' knowledge, no prior studies have looked at the effect of H2 receptor antagonists on the microbiome in healthy, full term infants.

ELIGIBILITY:
Inclusion Criteria:

* Full term, at least 2 months of age
* No exposure OR at least 14 days of exposure to H2-receptor antagonist medication
* No exposure to probiotics or antibiotics

Exclusion Criteria:

* Current or recent (within the past 14 days) gastrointestinal infection (viral, bacterial, or fungal)
* Gastrointestinal mucosal disease, or have clinically significant constipation
* Any history of exposure to proton pump inhibitors
* Unvaccinated infants
* Infants with weight-for-length either below the 3rd percentile for age or above the 97th percentile for age
* Infants with rapid weight gain, defined as change in weight-for-length z-score exceeding +0.67 from birth to 4 months of age or birth to 6 months of age

Ages: 2 Months to 12 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Infants must be healthy, male or female term infants (gestational age ≥37 weeks) who are at least 2 months old, on or off H2RA medication, who meet inclusion/exclusion criteria. Infants will be recruited from Nemours Children's Clinic and through local advertisements in the greater Wilmington / Northern Delaware area.
Sampling Method: Non-Probability Sample
Enrollment: 12 (Actual)
Dates: Start 2018-08-13 (Actual); Primary Completion 2019-04-30 (Actual); Study Completion 2019-07-31 (Actual)

PRIMARY OUTCOMES:
Microbiome taxa | At time of sampling - once at enrollment
  16S Metagenomic taxonomy of gut microbiome

CONTACTS AND LOCATIONS:
Overall Officials: Matthew Di Guglielmo, MD PhD, Principal Investigator — Nemours
Locations (1):
- Alfred I. duPont Hospital for Children, Wilmington, Delaware, United States

IPD SHARING:
Plan to Share IPD: Yes
16S metagenomic sequence data, deidentified, will be made available through either the database of Genotypes and Phenotypes (dbGap) or Sequence Read Archive (SRA).
Supporting Information: Analytic Code
Time Frame: At conclusion of the study.
Access Criteria: To be determined.